CLINICAL TRIAL: NCT04482140
Title: Post Approval Study to Evaluate the Safety and Performance of GENTA-FOIL Resorb® for the Prevention of Tissue Adhesions in Hand Surgery
Brief Title: Post Approval Study to Evaluate the Safety and Performance of GENTA-FOIL Resorb® in Hand Surgery
Status: Terminated | Type: Observational
Why Stopped: slow recruitment.
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); KAT General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 001GF
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Tissue Adhesions, Surgery-Induced
Keywords: Hand Mobility, Wound Healing, Functional restoration
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genta-Foil resorb®: Genta-Foil resorb® is a transparent collagen foil that forms a temporary barrier between the functional structures during the critical phase of wound healing. As a result, the ability of the tissue layers to slide against each other is retained. The absorbability of equine collagen means the foil can be left in place and does not require removal. The addition of the antibiotic Gentamicin is for self-protection since collagen implants are prone to bacterial contamination.
  Interventions: Device: Genta-Foil resorb®

INTERVENTIONS:
Device: Genta-Foil resorb® — Use of Genta-Foil resorb® to prevent adhesions in patients undergoing hand surgery

SUMMARY:
Single arm study to evaluate the safety and performance of Genta-Foil resorb® for the prevention of tissue adhesions

DETAILED DESCRIPTION:
GENTA-FOIL resorb® is an implantable, absorbable collagen barrier foil, which forms a temporary barrier between the functional structures during the critical phase of wound healing. As a result, the ability of the tissue layers to slide against each other is retained.

The objective of hand surgery is to promote wound repair, and regeneration of all motor and sensory functions of the hand and to restore the subject's hand mobility, and improve their quality of life. However, hand trauma and operations often lead to the formation of adhesions between the various tissue layers of the hand (e.g. muscles, tendons and nerves). Even with minimally invasive procedures and optimal aftercare, development of adhesions in the suture and wound areas is often unavoidable. Adhesion formation between repaired tendons and the surrounding tissue has been thought to be one of the most important factors that disturbs functional restoration. It is estimated that the adhesion, which can cause significant disability, occurs in about 30% of cases.

The purpose of this study is to investigate the use of GENTA-FOIL resorb® for the prevention of tissue adhesions measured by restoration in digital function in subjects undergoing hand surgery. The functional outcome of tendon injury after a repair depends on multiple factors such as age, injury level and type, type of repair, and post repair therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, ≥18 years of age;
2. Subject is willing and able to give written informed consent;
3. Subject is scheduled for one if the following surgical procedures:

   * 3a. extensor tendon repair zones I to VI.
   * 3b. flexor tendon repair zones I to VI.
   * 3c. open reduction and internal fixation to repair hand fractures of proximal phalanx, and/or middle phalanx, and/or metacarpals
4. Subject is willing and able to comply with the study procedures during surgery and the post-surgical follow up period.

Exclusion Criteria:

1. Subject is known to be sensitive to any of the device components e.g. Gentamicin (aminoglycosides) or equine collagen.
2. Subject is known to be non-compliant with medical treatment.
3. Subject has any known impaired renal function/autoimmune illness/neuromuscular disease (such as Parkinson's or Myasthenia Gravis).
4. Subject is currently taking an Aminoglycoside antibiotic as stand-alone treatment or in combination with other antibiotics
5. Subject is pregnant or actively breastfeeding.
6. Subject has active infection at surgical site
7. Subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with their ability to participate in the study, or affect the study outcomes.
8. Subject is currently enrolled in another clinical study that would interfere with their ability to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are undergoing hand surgery with the Genta-Foil resorb® device, and who meet all inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Restoration of hand mobility | At 90 days post-surgery
  Restoration of hand mobility will be assessed using functional assessment scoring Total Active Motion (TAM) at 90 days post-surgery. This will be measured by the modified Strickland scoring criteria. The success criteria is defined as TAM score of 75% or above at 90 days post-surgery. Restriction of TAM post-surgery is indicative of tissue adhesions, therefore this measure will demonstrate presence / absence of of tissue adhesions.

SECONDARY OUTCOMES:
Incidence of device related infections at surgical site up to 30 days post-surgery. | Up to 30 days post-surgery
  As per local Standard of Care wound assessment, absence or presence of wound signs infection will be recorded.
Incidence of device related adverse events | Up to 90 days post-surgery
  Evaluation of safety of GENTA-FOIL resorb® by recording of any device or procedure-related adverse events throughout the surgery during the follow-up period (day of surgery, at 7 days, 14 days, 30 days and 90 days post-surgery)
Subjective assessment of symptoms and abilities to perform activities by 90 days post-surgery | At 90 days post-surgery
  Study subjects requested to self assess symptoms and abilities to perform activities by 90 days post-surgery. Subjects will be asked to complete the standardised QuickDASH upper extremity outcome measure questionnaire. QuickDASH Outcome Measure tool measures the individual's ability to complete tasks at home and severity of symptoms. The tool uses 11 questions and a 5-point Likert Scale from which the patient can select an appropriate number corresponding to their severity / function level.
Wound healing without complications up to 30 days post-surgery. | Up to 30 days
  Standard of Care wound assessments will be performed at follow-up visits at day 7, day 14 and day 30 as appropriate, by a designated member of the Hand Dressing Clinic as per local Outpatient Wound Assessment Tool. As part of wound assessment, date of when wound is healed will be recorded during appropriate follow-up visit.
Change in patient pain scores (assessed using VAS) up to 90 days post-surgery. | Up to 90 days post-surgery
  Severity of localised pain in the affected hand or finger(s) will be measured using a Visual Analogue Scale (VAS). The VAS will be a 10cm horizontal line, with descriptors at each end [no pain (0cm), and worst imaginable pain (10cm)]. Subjects will be asked to place a mark on the scale that corresponds to their pain. The distance from the lower end of the scale will be measured and recorded.
Clinicians' satisfaction with the device at time of surgery | Immediately post-surgery
  Assessment of satisfaction with device conformability and ease of use. Assessed using a Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lipscombe, Principal Investigator — Whiston Hospital Mersey and West Lancashire Teaching Hospitals NHS Trust, Warrington Rd, Rainhill, Prescot
Locations (3):
- KAT Attica General Hospital, Athens, Athens, Greece
- United Kingdom (2):
  - Whiston Hospital - Mersey and West Lancashire Teaching Hospitals Trust, Rainhill, Merseyside
  - Royal Victoria Infirmary Newcastle Upon Tyne NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No